CLINICAL TRIAL: NCT03354195
Title: Comparative Clinical Outcomes and Function Study Between MAKO Robotic-Arm Assisted UKA in ACL Intact and Deficient Knees
Brief Title: MAKO-Uni-Knee Arthroplasty Clinical Outcomes and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-MAKO-001
Record Dates: First submitted 2017-10-20; First posted 2017-11-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Clinical Outcomes
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: During surgery, the ACL will be inspected, manually stressed and probed following standard techniques to assess its structure and function.(20, 21) The state of the ACL will be recorded and classified into one of four categories per these intra-operative examinations (22) and available pre-operative MRI data:
  Group 1 - intact ACL ligament
  Group 2 - intact but fibrillated (frayed) ligament)
  Group 3 - nearly completely torn ligament (>50% and disrupted)
  Assessment will be performed by the PI. Knees with ACLs classified as Group 1 and Group 2 will be accepted as functionally intact. Those classified as Group 3 will be deemed as having functionally absent ACLs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Group 1 - intact ACL ligament will be accepted as functionally intact
  unicompartmental knee arthroplasty with the Mako Robotic Arm-assisted system.
  Interventions: Procedure: Unicompartmental knee arthroplasty with the Mako Robotic Arm-assisted system.
- Group 2 (Active Comparator): Group 2 - intact but fibrillated (frayed) ligament) will be accepted as functionally intact
  unicompartmental knee arthroplasty with the Mako Robotic Arm-assisted system.
  Interventions: Procedure: Unicompartmental knee arthroplasty with the Mako Robotic Arm-assisted system.
- Group 3 (Active Comparator): Group 3 - nearly completely torn ligament (>50% and disrupted) will be deemed as having functionally absent ACLs
  unicompartmental knee arthroplasty with the Mako Robotic Arm-assisted system.
  Interventions: Procedure: Unicompartmental knee arthroplasty with the Mako Robotic Arm-assisted system.

INTERVENTIONS:
Procedure: Unicompartmental knee arthroplasty with the Mako Robotic Arm-assisted system. — All patients will receive the RESTORIS MCK (Multicompartmental Knee) Implant System, which is approved for use in unicompartmental knee arthroplasty with the Mako Robotic Arm-assisted system. The femoral component is constructed from cobalt chrome (CoCr) and the tibial component is constructed from an ultra-high molecular weight polyethylene (UHMWPE) insert and titanium (Ti) baseplate. UKA will be facilitated with MAKO Robotic-Arm Assisted Surgery, which has been shown in prior studies to lower pain and result in more accurate implant placement than manual UKA in a randomized controlled trial.(15)
  Other Names: UKA with Mako Robotic Arm-assisted system

SUMMARY:
This study represents a single-surgeon/institution, non-randomized, consecutive series, prospective and comparative cohort design. The Principal Investigator is anticipating 100 study patients in the INTACT group and 35 patients in the Anterior Cruciate Ligament-Deficient group.The schedule of events lists the imaging procedures and questionnaires to be completed at each visit.

Subjects will be consented and enrolled within 28 days prior to surgery and participate in follow-up visits for two years following their Unicompartmental Knee Arthroplasty. A 3-year enrollment duration is anticipated to enroll a minimum and consecutive series of 25 patients in the experimental Anterior Cruciate Ligament-deficient group. Over the same enrollment duration, 100+ patients with intact Anterior Cruciate Ligaments are expected to be in the control group and undergo Unicompartmental Knee Arthroplasty. The enrollment duration (3 years) and total study duration (5 years) are based on patient volume estimates provided by the Principal Investigator.

DETAILED DESCRIPTION:
To compare functional and clinical outcomes in patients with and without intact Anterior Cruciate Ligament undergoing uni-compartmental knee arthroplasty with MAKOplasty Robotic-Arm Assisted Surgery. The primary outcome measurement tools utilized will be the Knee Society Score (KSS) and Knee Injury and Osteoarthritis Outcomes Score (KOOS,JR). Both the Knee Society Score and Knee Injury and Osteoarthritis Outcomes Score (KOOS,JR) are validated scoring systems. Patient-reported outcome data will be collected at the following study time points:

* Preoperatively - Knee Society Score: Pre-Op, Knee Injury and Osteoarthritis Outcomes Score
* 3 weeks (±1 week) - Knee Society Score: Post-Operative, Knee Injury and Osteoarthritis Outcomes Score , Subject Global Satisfaction Survey
* 6 weeks (± 1 week) - Knee Society Score: Post-Operative, Knee Injury and Osteoarthritis Outcomes Score, Subject Global Satisfaction Survey
* 3 months (± 2 weeks) - Knee Society Score: Post-Operative, Knee Injury and Osteoarthritis Outcomes Score, Subject Global Satisfaction Survey
* 1 year (± 1 month) - Knee Society Score: Post-Operative, Knee Injury and Osteoarthritis Outcomes Score, Subject Global Satisfaction Survey
* 2 years (± 2 months) - Knee Society Score: Post-Operative, Knee Injury and Osteoarthritis Outcomes Score, Subject Global Satisfaction Survey

Subject Identification

Each subject will be assigned a unique subject number. Subject numbers will not be re-assigned or re-used for any reason. Only assigned subject numbers and associated subject age, Anterior Cruciate Ligament integrity classification, pre/intra-operative imagery information, and temporal outcome data will be shared with Sponsor. Only subjects who meet the inclusion/exclusion criteria and sign the Inform Consent Form will be assigned a unique study identification number.

Pre-Operative Anterior Cruciate Ligament Integrity

The structural integrity of the Anterior Cruciate Ligament will be determined clinically and pre-operatively with the following:

1. Lachman's anterior drawer test: Performed while the patient is in the supine position with the knee in 20° of flexion. The distal femur is fixed with one hand, while the other hand holds the proximal tibia with the thumb on the anteromedial joint line. The tibia is pulled ventrally, and the examiner estimates the ventral displacement of the tibia with respect to the femur. There are three possible outcomes: graded as 1+ (0-5 mm of displacement), 2+ (6-10 mm of displacement) or 3+ (greater than 10 mm of displacement) A 2+ or 3+ Lachman's test grade will be indicative of ACL instability.
2. Anterior drawer test: Performed with the patient in the supine position with the hips flexed to 45°, the knees flexed to 90° and the feet flat on the table. The thumbs are placed along the joint line on either side of the patellar tendon and the tibia is drawn forward anteriorly. An increased amount of anterior tibial translation compared with the opposite limb or lack of a firm end point may be indicative of either a sprain of the anteromedial bundle or complete tear of the Anterior Cruciate Ligament. If the tibia pulls forward or backward more than normal, the test is considered positive.
3. Pivot-Shift Test: Test is performed with the patient lying in supine position with the hip passively flexed to 30°.The examiner stands lateral to the patient on the side of the knee that is being examined. The lower leg and ankle is grasped maintaining 20 degrees of internal tibial rotation. The knee is allowed to sag into complete extension. The opposite hand grasps the lateral portion of the leg at the level of the superior tibiofibular joint, increasing the force of internal rotation. While maintaining internal rotation, a valgus force is applied to the knee while it is slowly flexed. If the tibia's position on the femur reduces as the knee is flexed in the range of 30 to 40 degrees or if there is an anterior subluxation felt during extension the test is positive for instability.
4. Biodex knee laxity test: This quantitative evaluation of knee laxity will be performed in accordance with the standardized procedures utilized by the Department of Physical Therapy at Florida Orthopaedic Institute.

Plain X-Ray

Knee osteoarthritis will be diagnosed and subjectively graded by taking plain radiographs in accordance with the Principal Investigator's Standard of Care, which include a (1) weight-bearing (WB) postero-anterior (PA) view, (2) sunrise view, and (3) lateral view. Degenerative disease of the knees will be graded per the Ahlback - Grades 1-5, increasing in severity or Kellgren and Lawrence Grade 0-4, increasing in severity classification systems. The Principal Investigator also uses a subjective classification system of mild, moderate, or severe osteoarthritis, which is captured in the clinic note.

Magnetic Resonance Imaging

A standardized imaging protocol will be utilized for all Magnetic Resonance Imaging images. Specifically, a 3D-proton density non-fat suppressed fast spin echo sequence shall be used. Magnetic Resonance Imaging of the knee will be obtained prior to surgery using the parameters as requested by the Sponsor using Florida Orthopaedic Institute Siemens Aera 1.5T Magnetic Resonance Imaging scanner: TR/TE=1000/46, Flip angle=120°, repetition time=1000msec, echo time=46msec, bandwidth=97.3 Hz/pixel, matrix size= 320x300 pixels. The Sponsor has requested the use of a 3T magnet, but Florida Orthopaedic Institute currently has 1.5T magnets in their Magnetic Resonance Imaging scanners, so this request cannot be accommodated. We will perform a scan with the 1.5T magnet and share with Sponsor to confirm that the available imagery information is acceptable for their purposes.

Computed Tomography (CT) Scans

A Computed Tomography scan of the knee will be obtained prior to surgery using the standardized partial knee arthroplasty Computed Tomography scanning protocol with bone mineral density (BMD) phantom protocol as provided by the Sponsor. Sponsor will provide the phantom for use during scanning. A pre-operative Computed Tomography scan is required as the Standard of Care for robotic-arm assisted knee procedures. Each patient's Computed Tomography scan is used to create a 3D model of the patient's anatomy for accurate implant planning, bone resection and implant placement.

KOOS-JR

The abbreviated version of the Knee Injury and Osteoarthritis Outcome Score (KOOS) survey is a validated and self-reported questionnaire (7 questions) designed to measure "knee health" as it reflects aspects of pain, symptom severity, and activities of daily living (ADL) including movement or activities that are directly relevant and difficult for patients with knee Osteoarthritis.The Knee Injury- Osteoarthritis Outcomes Score-JR knee survey consists of 7 questions pertaining to knee stiffness, knee pain, and physical function. The survey will be administered to all patients at baseline, 3 weeks, 6 weeks, 3 months, 1 year and 2 years.

KSS

The knee society score has been in use for over 20 years and is a simple, objective means to measure a patient's functional ability before and after surgery (11-13). It includes ROM assessment. The Principal Investigator will utilize the updated Knee Society Score (2011), which has been modified to include both an objective physician-derived component with a subjective patient-derived component that evaluates pain relief, functional abilities, satisfaction, and fulfillment of expectations. This updated scoring system prioritizes the patient perspective, to better track patient expectations, satisfaction, and activity levels than was possible with its predecessor. Patients will complete this survey with the Principal Investigator at all study time points.

Global Satisfaction Survey

This custom, 2-page survey has been designed by the study team to track patient satisfaction after their Unicompartmental Knee Arthroplasty over time. It's a simple, seven-item survey that also includes a Visual Analogue Scale for knee pain. The survey will be administered to all patients at all post-operative visits.

Intra-Operative Anterior Cruciate Ligament Integrity

During surgery, the Anterior Cruciate Ligament will be inspected, manually stressed and probed following standard techniques to assess its structure and function.The state of the Anterior Cruciate Ligament will be recorded and classified into one of four categories per these intra-operative examinations and available pre-operative Magnetic Resonance Imaging data:

Group 1 - intact Anterior Cruciate Ligament Group 2 - intact but fibrillated (frayed) ligament) Group 3 - nearly completely torn ligament (>50% and disrupted)

Assessment will be performed by the Principal Investigator. Knees with Anterior Cruciate Ligaments classified as Group 1 and Group 2 will be accepted as functionally intact. Those classified as Group 3 will be deemed as having functionally absent Anterior Cruciate Ligaments.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet these criteria to participate in this study:

1. Patients with isolated, symptomatic femorotibial knee arthritis and candidates for UKA;
2. Patients ≥ 21 years old;
3. Patients with intact and non-functional ACLs as determined through pre-operative imaging, knee laxity tests, rotational stability tests, and intraoperative ACL classification;
4. Patients willing and able to sign an informed consent;
5. Patients willing and able to comply with 2-year follow-up commitments.

Exclusion Criteria:

Any subject who meets any of the exclusion criteria will be excluded from participation in this study:

1. Patients with RA;
2. Patients with BMI >40;
3. Patients with ROM arc > 75°;
4. Patients with greater than 10º of hyperextension;
5. Patients with greater than 15º of varus or valgus deformity;
6. Patients with active infection;
7. Patients without sufficient bone stock to allow appropriate insertion and fixation of the prosthesis;
8. Patients without sufficient soft tissue integrity to provide adequate stability;
9. Patients with either mental or neuromuscular disorders that do not allow control of the knee joint;
10. Patients whose weight, age or activity level might cause extreme loads and early failure of the system.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Functional and Clinical Outcomes comparing patients with and without intact Anterior Cruciate Ligaments undergoing arthroplasty with MAKO Robotic-Arm Assisted Surgery. | Baseline (screening), compared to a 24 month follow-up visit. There are also several additional time points from 3 weeks, 6 weeks, 3 months, 6 months and 12 months where the functional and clinical outcomes are assessed.
  Knee Society Score (KSS) and Knee Injury and Osteoarthritis Outcome Score (KOOS)

SECONDARY OUTCOMES:
Height and Weight | Baseline (screening)
  to calculate subjects BMI
Computed Tomography | Baseline (screening)
  A pre-operative CT scan is required as the Standard of Care for robotic-arm assisted knee procedures.
Magnetic Resonance Imaging | Baseline (screening)
  MRI of the knee will be obtained prior to surgery using the parameters as requested by the Sponsor
Radiographs (3 views) | Baseline (screening)
  Knee osteoarthritis will be diagnosed and subjectively graded by taking plain radiographs in accordance with the PI's Standard of Care, which include a (1) weight-bearing (WB) postero-anterior (PA) view, (2) sunrise view, and (3) lateral view. Degenerative disease of the knees will be graded per the Ahlback Grades 1-5, increasing in severity or Kellgren and Lawrence ,Grade 0-4, increasing in severity classification systems. The Principal Investigator also uses a subjective classification system of mild, moderate, or severe osteoarthritis, which is captured in the clinic note.
Global Satisfaction Survey | Baseline (screening), 3 weeks, 6 weeks, 3 months, 12 months, 24 months
  2-page survey has been designed by the study team to track patient satisfaction after their UKA over time
Intra-Operative ACL Integrity | Enrollment (procedure day)
  Knees with ACLs classified as Group 1 and Group 2 will be accepted as functionally intact. Those classified as Group 3 will be deemed as having functionally absent ACLs.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make the IPD available.